CLINICAL TRIAL: NCT01359306
Title: Right Ventricular Damage in ST-Elevation Myocardial Infarction. Risk Stratification by Visualization of Wall Motion, Edema and Delayed Enhancement Cardiovascular Magnetic Resonance
Brief Title: Right Ventricular Damage in Cardiovascular Magnetic Resonance
Status: Completed | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Matthias Grothoff MD, University Leipzig Heart Center
Other Study IDs: RV-Damage 1/2007
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Right ventricular infarction; Cardiovascular Magnetic Resonance; Prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum for assessment of creatine kinase myocardial band
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the predictors of right ventricular damage (RVD) assessed by wall motion abnormalities, edema, myocardial salvage and delayed enhancement (DE)cardiac magnetic resonance imaging in acute ST-elevation myocardial infarction (STEMI) and its prognostic significance.

The investigators hypothesize that ischemia related changes of the myocardium are also visible in the right ventricle and that they have an impact on patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Onset of symptoms <12 h before angioplasty.
* ST-segment elevation of at least 0.1 mV in ≥2 extremity leads or at least 0.2 mV in ≥2 precordial leads.

Exclusion Criteria:

* Contraindications to CMR as implanted defibrillators, pacemakers, ferromagnetic intracranial metallic implants or pulmonary metallic splints and claustrophobia. A further exclusion criterion was prior fibrinolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 524 consecutive patients with ST elevation myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2006-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Event | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Grothoff, MD, Principal Investigator — Heart Center Leipzig - University Hospital

REFERENCES:
- [Derived] Grothoff M, Elpert C, Hoffmann J, Zachrau J, Lehmkuhl L, de Waha S, Desch S, Eitel I, Mende M, Thiele H, Gutberlet M. Right ventricular injury in ST-elevation myocardial infarction: risk stratification by visualization of wall motion, edema, and delayed-enhancement cardiac magnetic resonance. Circ Cardiovasc Imaging. 2012 Jan;5(1):60-8. doi: 10.1161/CIRCIMAGING.111.967810. Epub 2011 Nov 11. PMID 22080332